CLINICAL TRIAL: NCT04704700
Title: Evaluate the Rotator Cuff Repair With "InSpace" VS Without "InSpace"
Acronym: ESPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Bizet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A02443-36
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Repair of a Cuff Tear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with inspace device (Active Comparator)
  Interventions: Device: repair of a cuff tear
- patient without inspace device (Placebo Comparator)
  Interventions: Device: repair of a cuff tear

INTERVENTIONS:
Device: repair of a cuff tear — Group (Treatment): Arthroscopic Implantation of the System InSpace on a repaired rotator cuff tendon
  Arms: patient with inspace device
Device: repair of a cuff tear — Group (Control): standard Arthroscopic repair of the cuff rotator
  Arms: patient without inspace device

SUMMARY:
Evaluate the re-rupture rate 12 months following the intervention in a group with and a group without a spacer

ELIGIBILITY:
Inclusion Criteria:

* First intention of the rotator cuff
* Repairable supraspinatus and infraspinatus type 2 rupture (according to the PATTE classification, tendon retraction at the top of the humeral head)
* No surgical history
* Patient who has given his participation agreement to participate in the observational study after information by the surgeon,
* Patient living in France and having the capacity to answer alone to the survey.
* Subject affiliated to a social security scheme
* Lack of participation in another clinical study

Exclusion Criteria:

* Major subject protected by law, under curatorship or tutorship
* Known allergy to Inspace medical device materials (PLA and -θ-caprolactone copolymer)
* Osteoporosis
* Damaged cartilage
* Isolated rupture of the suprascapularis
* Glenohumeral instability
* Pseudo-paralytic shoulder- Infection
* Necrosis
* Major joint trauma
* Pregnant or breastfeeding women

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the re-rupture rate | 12 months
  with radiological imaging

SECONDARY OUTCOMES:
Evaluate mobility | up to 12 months
  the Constant score
Assess shoulder pain | up to 12 months
  VISUAL ANALOGIC SCALE
the quality of life assessed | up to 12 months
  Simple Shoulder Test, Subjective Shoulder Value and American Shoulder and Elbow Surgeons Shoulder Score
resumption of work | up to 12 months
  Physicians Global Assessment for resumption of work

CONTACTS AND LOCATIONS:
Overall Officials: philippe VALENTI, DOCTOR, Principal Investigator — Clinique Bizet
Locations (1):
- Clinique Bizet, Paris, France